CLINICAL TRIAL: NCT03738163
Title: A Prospective Post Market Clinical Follow-up Investigation With Epaderm® Cream to Confirm Performance and Safety Parameters
Brief Title: A Clinical Investigation With Epaderm® Cream
Acronym: PD-539878
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Epaderm01
Record Dates: First submitted 2018-10-26; First posted 2018-11-13 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Eczema; Psoriasis; Dry Skin; Eczema
MeSH Terms: conditions — Eczema; Psoriasis

STUDY DESIGN:
Intervention Model Description: infants (0-36 months old), children (3-18 years old) and adults (>18 years old)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epaderm Cream (Other): This is an open, non randomised single arm study.
  Interventions: Device: Epaderm Cream

INTERVENTIONS:
Device: Epaderm Cream — The treatment with the investigational device will be according to the prescription by the investigator together with the instruction stated on the investigational device.

SUMMARY:
This investigation is designed as a prospective, non-randomised, single arm clinical investigation. Data is collected from approximately 120 evaluable subjects, divided into three groups of approximately 40 subjects; infants (0-36 months old), children (3-18 years old) and adults (>18 years old), with the following indications: eczema, psoriasis and other dry skin conditions. Each subject will be followed during 4 weeks treatment, with a visit at baseline (visit 1), at 2 weeks (visit 2) and at 4 weeks (visit 3) treatment.

DETAILED DESCRIPTION:
Primary Endpoint Skin hydration after treatment with Epaderm Cream up to 4 weeks, evaluated by the subject using a questionnaire.

Secondary Endpoints

1. Skin hydration after treatment with Epaderm Cream up to 4 weeks, evaluated by investigator/nurse using a questionnaire.
2. Skin hydration after treatment with Epaderm Cream up to 4 weeks, using a non-invasive device MoistureMeterEpiD.
3. Investigator/nurse evaluation of skin softness after 2 and 4 weeks treatment, using a questionnaire.
4. Subject evaluation of skin softness after 2 and 4 weeks treatment, using a questionnaire.
5. Investigator/nurse evaluation regarding:

   * Clinical signs/conditions of the affected skin and changes thereof
   * Did the product prolong the relapse period for flares?
6. Subject evaluation regarding:

   * Did you use Epaderm Cream according to prescription?
   * Comfort during treatment
   * Time of onset of effect
   * Did the product have the expected effect
   * Overall impression
   * Was the investigational device used as a skin cleanser?
7. Concomitant and previous medication and treatment
8. Number of Adverse Device Effects (ADEs) related to the use of Epaderm Cream during the investigation

ELIGIBILITY:
Inclusion Criteria:

1. Subjects suitable for treatment with Epaderm Cream, as deemed by the investigator and according to intended use (eczema, psoriasis and other dry skin conditions).
2. Subject or subject's legal representative must be able to read and sign the Patient Information and Consent Form.

Exclusion Criteria:

1. Known allergy/hypersensitivity to any of the components of Epaderm Cream.
2. Subject not suitable for the investigation according to the investigator's judgement.
3. Subject participating in other ongoing similar clinical studies or other clinical studies which could interfere with this investigation, as judged by the investigator.
4. Subject previously enrolled in the current clinical investigation.

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2020-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzannah August, MD, Principal Investigator — Poole Hospital
Locations (2):
- United Kingdom (2):
  - Poole Hospital NHS Foundation Trust, Poole, Dorset
  - Whiteladies Medical Group, Bristol

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Epaderm Cream
Started | 121
Completed | 114
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Epaderm Cream
Number analyzed (Participants) | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36
  Between 18 and 65 years | 44
  >=65 years | 41
Age, Continuous [Mean (Full Range); unit: years] | 30.5 [0.3 to 90]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 7 subjects withdrew from the study.
  Participants
    number analyzed (Participants) | 114
    Female | 51
    Male | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 121

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improved Skin Moisturization
Description: Participants were considered to have improved moisturization if they responded strongly agree or agree on the questionnaire. Evaluations were carried out in the same affected spot from a scale of Strongly agree, Agree, Neither agree nor disagree,
  Disagree, Strongly disagree where Strongly agree is the most improved skin moisturization:
Time Frame: Assessed at 2 weeks and 4 weeks visit, 4 weeks visit reported
Measure: Count of Participants; unit: Participants
Arm/Group | Epaderm Cream
Number analyzed (Participants) | 121
Participants | 114

2. Secondary Outcome: Number of Participants With Improved Skin Softness
Description: Participants were considered to have improved softness if they responded strongly agree or agree on the questionnaire. Evaluations were carried out in the same affected spot from a scale of Strongly agree, Agree, Neither agree nor disagree, Disagree, Strongly disagree where Strongly agree is the most improved skin softness.
Time Frame: Assessed at 2 weeks and 4 weeks visit, 4 weeks visit reported
Measure: Count of Participants; unit: Participants
Arm/Group | Epaderm Cream
Number analyzed (Participants) | 114
Participants | 82

3. Secondary Outcome: Number of Participants With Improved Overall Dry Skin/Xerosis
Description: Participants were considered to have improved overall dry skin if they responded 'absent' or 'faint scaling' on the questionnaire. Evaluations were carried out in the same affected spot from a scale of 0= Absent, 1= Faint scaling, faint roughness and dull appearance, 2= Small scales in combination with a few larger scales, slight roughness, whitish appearance, 3= Small and larger scales uniformly distributed, definite roughness, possibly slight redness and possibly a few superficial cracks, 4= Dominated by large scales, advanced roughness, redness present, eczematous changes and cracks where 'absent' or 'fanit scaling' refers to improved overall dry skin.
Time Frame: Assessed at 2 weeks and 4 weeks visit, 4 weeks visit reported
Measure: Count of Participants; unit: Participants
Arm/Group | Epaderm Cream
Number analyzed (Participants) | 114
Participants | 100

4. Secondary Outcome: Number of Participants Who Confirmed Overall Effect and Comfort of Treatment
Description: Participants confirmed the comfort during treatment from a scale of Very Poor, Poor, Average, Good and Excellent where Excellent is considered the most comforting during treatment.
Time Frame: Assessed at 2 weeks and 4 weeks visit, 4 weeks visit reported
Measure: Number; unit: participants
Arm/Group | Epaderm Cream
Number analyzed (Participants) | 114
participants | 101

5. Secondary Outcome: Number of Participants With Adverse Device Effects (ADEs)
Description: Number of Adverse Device Effects (ADEs) related to the use of Epaderm Cream during the investigation.
Time Frame: Evaluated at every follow-up visit (2 weeks and 4 weeks visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Epaderm Cream
Number analyzed (Participants) | 114
Participants | 10

6. Secondary Outcome: Number of Participants Who Reported Applying Epaderm Cream Twice a Day
Description: Frequency of Epaderm Cream application. Participants were asked how often Epaderm Cream was applied either once a day, twice a day, three times a day or four times a day with twice a day application being the most frequent.
Time Frame: Assessed at 2 weeks and 4 weeks visit, 4 weeks visit reported
Measure: Count of Participants; unit: Participants
Arm/Group | Epaderm Cream
Number analyzed (Participants) | 114
Participants | 67

7. Secondary Outcome: Number of Participants With Improvement of Skin Moisturization By Week 4
Description: Participants confirmed the time to visualize improvement of skin moisturization from the range immediately, within 2 weeks or not at all where immediately refers to the most increased improvements seen.
Time Frame: Assessed at 2 weeks and 4 weeks visit. Improvement within 4 weeks visit reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Epaderm Cream
Number analyzed (Participants) | 114
Participants | 107

8. Secondary Outcome: Number of Participants Who Used Epaderm as a Skin Cleanser
Description: Participants were asked to confirm if the product was used as a skin cleanser by answering yes or no where yes confirmed use of Epaderm cream as a skin cleanser.
Time Frame: Assessed at 2 weeks and 4 weeks visit, 4 weeks visit reported where participates answered 'yes'.
Measure: Count of Participants; unit: Participants
Arm/Group | Epaderm Cream
Number analyzed (Participants) | 114
Participants | 75

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a period of 4 weeks from the baseline visit to the final follow-up visit.
Arm/Group | Epaderm Cream
All-Cause Mortality (participants affected / at risk) | 0/121
Serious Adverse Events (participants affected / at risk) | 0/121
Other Adverse Events (participants affected / at risk) | 10/121
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epaderm Cream (N=121)
Flare of eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Intermittent rash (Skin and subcutaneous tissue disorders) | 4 (4) — Redness & itch
Inflammatory reaction (Skin and subcutaneous tissue disorders) | 2 (2)
Worsening of the skin (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT03738163/Prot_SAP_000.pdf